CLINICAL TRIAL: NCT06934382
Title: A Phase 1 Study of Allogeneic Anti-CD7 CAR-T Cells (BEAM-201) in Relapsed/Refractory T-cell Acute Lymphoblastic Leukemia (T-ALL) or T-cell Lymphoblastic Lymphoma (T-LLy)
Brief Title: Anti-CD7 CAR-T Cells in Relapsed/Refractory T-Cell Acute Lymphoblastic Leukemia or Lymphoma
Acronym: 24CT015
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Collaborators: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Chief, Cell Therapy and Transplant Section Director, Susan S. and Stephen P. Kelly Center for Cancer Immunotherapy Medical Director, Cell and Gene Therapy Lab, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24CT015, 25-023121, BTX-ALT-00
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: T-Cell Acute Lymphoblastic Leukemia/Lymphoma
Keywords: CART; T-cell leukemia; T-cell lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Leukemia, T-Cell; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Arm (Experimental): The dose escalation portion of the trial will use a standard "3+3" design to establish the recommended maximum tolerated dose of BEAM-201 cells. Three dose escalations of BEAM-201 are planned for the dose escalation phase, with one dose de-escalation level if needed.
  Interventions: Biological: Allogeneic anti-CD7 CAR-T cells (BEAM-201)
- Dose Expansion Arm (Experimental): If at least one dose level of the dose escalation phase is determined to be safe, the dose expansion phase of the trial will be opened to enrollment.
  Interventions: Biological: Allogeneic anti-CD7 CAR-T cells (BEAM-201)

INTERVENTIONS:
Biological: Allogeneic anti-CD7 CAR-T cells (BEAM-201) — The investigational agent in this protocol is allogeneic anti-CD7 CART cells (BEAM-201). BEAM-201 is comprised of allogeneic anti-CD7 CAR-T cells edited by 4 gRNAs and a single mRNA encoding a CBE, then transduced with a lentiviral vector (LVV) encoding the anti-CD7 chimeric antigen receptor (CAR) molecule.
  Other Names: BEAM-201

SUMMARY:
This will be a Phase 1, open-label study to evaluate the safety and efficacy of BEAM-201 in patients with R/R T-ALL or T-LLy. BEAM-201 is an allogeneic anti-CD7 CART therapy.

DETAILED DESCRIPTION:
Despite favorable outcomes in newly diagnosed patients, approximately 20% of pediatric and young adult T-ALL patients and 40% of adult patients will have refractory disease or will relapse within 2 years of their initial diagnosis. Survival rates of patients with relapsed disease remain below 35%. For recurrent disease, allogeneic hematopoietic stem cell transplant (HSCT) is the only known potentially curative treatment. However, a prerequisite to HSCT is obtaining a complete remission, which remains a significant challenge as only 40 to 50% of patients achieve a second remission with current reinduction regimens with salvage rates even lower for patients with disease that is refractory to first-line chemotherapy.

BEAM-201 is an allogeneic anti-CD7 CAR T cell product that has shown promising early evidence of efficacy, with 3 out of 4 adult T-ALL patients infused had a CRi/CR ≥28 days after infusion. Safety of BEAM-201 has been favorable and consistent with known adverse events associated with other CAR T cell therapies.

Given the current treatment landscape of T-ALL/T-LLy, promising clinical experience with BEAM-201, and that >98% of T-ALL cases highly and homogenously express CD7 protein on the surfaces of their lymphoblasts, the investigators think there is compelling rationale in further investigating the safety and efficacy of BEAM-201 in pediatric patients.

ELIGIBILITY:
Patients must meet all the following criteria to be eligible for enrollment into the study:

1. Patients (ages ≥ 18 years) or parent/legal guardians (for patients ages < 18 years) must provide signed, written informed consent according to local IRB and institutional requirements.
2. Ages 0 to 29 years.
3. T-ALL/T-LLy in second or greater relapse, first relapse post-transplant, or chemotherapy-refractory disease. Specifically:

   1. Second or greater relapse or post-transplant relapse, defined as:

      * BM with ≥ 5% lymphoblasts by morphologic assessment or evidence of extramedullary disease after second documented CR; OR
      * Flow cytometric confirmation of relapsed T-ALL of at least 0.1% after second CR documented to have been MRD negative < 0.1%; OR
      * Any detectable relapsed disease post-allogeneic HSCT with flow cytometric confirmation of T-ALL of at least 0.1%; OR
      * Biopsy confirmed evidence of relapsed T-LLy after second CR; OR
      * Any detectable disease post-allogeneic transplant with biopsy confirmed evidence of T-LLy
   2. Refractory disease, defined as:

      * Primary refractory T-ALL or T-LLy, defined as failure to achieve CR after induction chemotherapy, per investigator assessment and based on biopsy-or MRD-confirmed evidence of residual T-ALL or T-LLy; OR
      * Relapsed, refractory disease, defined as > 0.1 % MRD or morphologic evidence of disease or evidence of residual T-LLy after 1 course of re-induction chemotherapy for patients who have relapsed after previously achieving a CR NOTE: Patients with mixed phenotype acute leukemia with T cell dominant phenotype may be enrolled if the aforementioned criteria are met.
4. Documentation of CD7 expression on leukemic or T-LLy blasts (defined as at least 90% of blasts positive for CD7 by flow cytometry or immunohistochemistry).
5. Patients with prior or current history of CNS3 disease will be eligible if CNS disease is responsive to therapy
6. Eligible for myeloablative conditioning for and allogeneic HSCT based on the investigator's assessment with an available donor identified by a FACT accredited transplant center.
7. Lansky Performance Status (ages < 16 years at time of consent) or Karnofsky Performance Status (KPS) (ages ≥ 16 years at time of consent) score of ≥ 50.
8. Patients of childbearing potential must have a negative urine or serum pregnancy test at screening.
9. Adequate organ function defined as:

   1. Adequate Serum creatinine based on age/gender
   2. ALT ≤ 5x ULN in the absence of ALL infiltration of the liver
   3. Bilirubin ≤ 3 × ULN for age Note: ALT and/or bilirubin results that exceed this range are acceptable if, in the opinion of the physician-investigator (or as confirmed by liver biopsy), the abnormalities are directly related to ALL infiltration of the liver.
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and <Grade 3 hypoxia; DLCO ≥40% (corrected for anemia if necessary) if PFTs are clinically appropriate as determined by the investigator.
   5. Cardiac echocardiography (ECHO) with left ventricular shortening fraction (LVSF) ≥ 30% or left ventricular ejection fraction (LVEF) ≥ 50%. In cases where quantitative assessment of LVSF/LVEF is not possible, a statement by the cardiologist that the ECHO shows qualitatively normal ventricular function will suffice
10. Patients who are sexually active and of reproductive potential must agree to use an acceptable form of highly effective contraception from consent to 12 months after BEAM 201 infusion.

4.2 Exclusion Criteria

Patients who meet any of the following criteria will be disqualified from entering the study:

1. Active hepatitis B or active hepatitis C
2. Active HTLV infection
3. HIV infection
4. Uncontrolled, active bacterial, viral, or fungal infection.
5. CNS disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
6. Clinically active CNS dysfunction or known history of irreversible central neurological toxicity related to prior antileukemic therapy.
7. Receipt of prior CD7 targeted therapy.
8. Radiation therapy within 2 weeks prior to completion of screening, other than prophylaxis for CNS disease.
9. Acute GVHD that is grade ≥ 2 and requiring systemic immunosuppression (corticosteroids), or chronic GVHD that is mild, moderate, or severe and requiring systemic immunosuppression (corticosteroids). Grade 1 acute GVHD not requiring immunosuppression is allowable.
10. Undergone HSCT within 90 days prior to completion of screening (or donor leukocyte infusion, if received within 30 days prior to completion of screening).
11. Any other condition that would make the patient ineligible for HSCT as determined by the investigator.
12. Known primary immunodeficiency or BM failure syndrome.
13. Atrial fibrillation/flutter (not including isolated episodes that responded to medical management)
14. Clinically significant pericardial effusion
15. Myocardial infarction within the last 12 months
16. QT interval corrected for heart rate > 480 msec
17. Cardiac dysfunction NYHA (New York Heart Association) III or IV
18. Patients with an autoimmune disorder requiring systemic immunosuppressive therapy that cannot be safely withheld for 3 months.

    Concurrent use of systemic corticosteroids for diagnoses unrelated to T-ALL/T-LLy is prohibited, with exception of physiologic corticosteroid replacement therapy treatment for adrenal insufficiency.
19. Pregnant or breastfeeding

Ages: 0 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerate Dose of Beam 201 Cells | 5 years
  The Maximum Tolerated Dose will be determined by measuring the incidence of dose limiting toxicities following administration of the product.
Frequency of Adverse Events Following Beam-201 administration | 5 years
  Frequency of Adverse events will be measured by evaluating the frequency and severity of treatment related adverse events following administration of Beam-201 Cells

SECONDARY OUTCOMES:
• Determine the overall response rate following BEAM-201 infusion | 5 years
  Defined as the frequency of patients who achieve complete remission or partial response following treatment with Beam 201
Determine depth of response based on MRD for patients with clinical responses following BEAM-201 infusion | 5 years
  Evaluated as the frequency of patients who have minimal residual disease through next generation sequencing
Determine the proportion of patients treated with BEAM-201 who are deemed appropriate for stem cell transplant | 5 years
  As evaluated the percentage of patients who proceed to stem cell transplant following Beam-201 administration
• Determine duration of response for patients with clinical responses following BEAM 201 infusion | 5 years
  Duration of Response will be measured by the average number of months in remission after Beam 201 administration
Determine overall survival following BEAM-201 infusion | 5 years
  Overall survival will be measured as proportion of subjects who remain alive 12 months after administration with Beam-201 cells

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Diorio, MD, Principal Investigator — Children's Hospital of Philadelphia; Stephan Grupp, MD, PhD, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No